CLINICAL TRIAL: NCT07171749
Title: Prevalence of Hemolytic Uremic Syndrome (HUS) in Pediatrics at Assiut University Children's Hospital: A Prospective Study
Brief Title: Prevalence of Hemolytic Uremic Syndrome (HUS) in Pediatrics
Status: Not yet recruiting | Type: Observational
Sponsor: Assiut University (Other)
Responsible Party: Principal Investigator, Hala Ali Abdelmawgoud Abd Elgied, Principal Investigator, Assiut University
Other Study IDs: Prevelance of HUS
Record Dates: First submitted 2025-09-06; First posted 2025-09-15 (Actual); Last update posted 2025-09-15 (Actual); Status verified 2025-09

CONDITIONS: Prevalence of Hemolytic Uremic Syndrome

STUDY DESIGN:
Observational Model: Other | Time Perspective: Cross-Sectional
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

SUMMARY:
To determine the prevalence of hemolytic uremic syndrome (HUS) among pediatric patients admitted to Assiut University Children's Hospital, and to describe the demographic, clinical, and laboratory characteristics of the affected population.

DETAILED DESCRIPTION:
Hemolytic uremic syndrome (HUS) is a rare but serious condition characterized by the triad of microangiopathic hemolytic anemia, thrombocytopenia, and acute kidney injury. [1] Two main subtypes of HUS are recognized. The majority of pediatric cases are classified as typical HUS, most frequently associated with Shiga toxin-producing Escherichia coli (STEC) infection. In contrast, atypical HUS (aHUS) is less common, accounting for approximately 5-10% of cases, and is linked to dysregulation of the complement system. The clinical course and prognosis differ significantly between these subtypes.[2].

Understanding the prevalence of HUS is critical for early recognition and timely intervention, especially in resource-limited settings. [3] Complications of HUS can be severe and include neurological manifestations, hypertension, persistent renal impairment, and in some cases, death. Early diagnosis and supportive care are critical for improved outcomes [4].

Local factors such as water safety, sanitation, access to early antibiotics, and public health surveillance greatly affect the observed prevalence. [5] The management of typical HUS caused by STEC is generally supportive. [6] For aHUS, early treatment is crucial to avoid end-stage renal disease (ESRD) and mortality. The cornerstones of treatment for aHUS are first-line therapy with eculizumab [7]

ELIGIBILITY:
Inclusion Criteria:

* Patients aged below 18 years at the time of diagnosis.
* Confirmed diagnosis of HUS based on the clinical triad (microangiopathic hemolytic anemia, thrombocytopenia, and acute kidney injury).

Exclusion Criteria:

* Patients aged 18 years or above at the time of diagnosis.
* Incomplete or missing medical records that do not confirm the diagnosis.

Ages: 1 Day to 18 Years | Sex: All
Age Groups: Child, Adult
Study Population: Pediatric patients (aged <18 years) who were diagnosed with hemolytic uremic syndrome (HUS) and admitted to Assiut University Children's Hospital during the period from 1 October 2025 to 30 September 2026.
Sampling Method: Non-Probability Sample
Enrollment: 50 (Estimated)
Dates: Start 2025-10-01 (Estimated); Primary Completion 2026-09-30 (Estimated); Study Completion 2026-10-30 (Estimated)

PRIMARY OUTCOMES:
Prevalence of Hemolytic Uremic Syndrome (HUS) among Pediatric Patients | Within 12months of enrollment (october 2025-September 2026)
  The proportion of pediatric patients diagnosed with HUS out of the total number of children admitted to Assiut University Children's Hospital during the study period. Diagnosis will be based on clinical, laboratory, and imaging criteria.

IPD SHARING:
Plan to Share IPD: Undecided

REFERENCES:
- [Result] Franchini M. Atypical hemolytic uremic syndrome: from diagnosis to treatment. Clin Chem Lab Med. 2015 Oct;53(11):1679-88. doi: 10.1515/cclm-2015-0024. PMID 25803082
- [Result] Joseph A, Cointe A, Mariani Kurkdjian P, Rafat C, Hertig A. Shiga Toxin-Associated Hemolytic Uremic Syndrome: A Narrative Review. Toxins (Basel). 2020 Jan 21;12(2):67. doi: 10.3390/toxins12020067. PMID 31973203
- [Result] Jenssen GR, Hovland E, Bjerre A, Bangstad HJ, Nygard K, Vold L. Incidence and etiology of hemolytic-uremic syndrome in children in Norway, 1999-2008--a retrospective study of hospital records to assess the sensitivity of surveillance. BMC Infect Dis. 2014 May 16;14:265. doi: 10.1186/1471-2334-14-265. PMID 24884396
- [Result] Yerigeri K, Kadatane S, Mongan K, Boyer O, Burke LLG, Sethi SK, Licht C, Raina R. Atypical Hemolytic-Uremic Syndrome: Genetic Basis, Clinical Manifestations, and a Multidisciplinary Approach to Management. J Multidiscip Healthc. 2023 Aug 4;16:2233-2249. doi: 10.2147/JMDH.S245620. eCollection 2023. PMID 37560408
- [Result] Zagozdzon I, Szczepanska M, Leszczynska B, Jarmuzek W, Miklaszewska M, Tkaczyk M, Medynska A, Wieczorkiewicz-Plaza A, Zachwieja J, Protas P, Rosinska P, Jacher U, Trembecka-Dubel E, Zwolinska D, Zurowska A. Changing Epidemiology and Outcomes of Hemolytic Uremic Syndrome in Children: A Prospective National Cohort Study from the Polish Pediatric HUS Registry and the Polish Registry of Renal Replacement Therapy in Children. J Clin Med. 2024 Oct 30;13(21):6499. doi: 10.3390/jcm13216499. PMID 39518638
- [Result] McKee RS, Schnadower D, Tarr PI, Xie J, Finkelstein Y, Desai N, Lane RD, Bergmann KR, Kaplan RL, Hariharan S, Cruz AT, Cohen DM, Dixon A, Ramgopal S, Rominger A, Powell EC, Kilgar J, Michelson KA, Beer D, Bitzan M, Pruitt CM, Yen K, Meckler GD, Plint AC, Bradin S, Abramo TJ, Gouin S, Kam AJ, Schuh A, Balamuth F, Hunley TE, Kanegaye JT, Jones NE, Avva U, Porter R, Fein DM, Louie JP, Freedman SB; Pediatric Emergency Medicine Collaborative Research Committee and Pediatric Emergency Research Canada. Predicting Hemolytic Uremic Syndrome and Renal Replacement Therapy in Shiga Toxin-producing Escherichia coli-infected Children. Clin Infect Dis. 2020 Apr 10;70(8):1643-1651. doi: 10.1093/cid/ciz432. PMID 31125419
- [Result] Bayer G, von Tokarski F, Thoreau B, Bauvois A, Barbet C, Cloarec S, Merieau E, Lachot S, Garot D, Bernard L, Gyan E, Perrotin F, Pouplard C, Maillot F, Gatault P, Sautenet B, Rusch E, Buchler M, Vigneau C, Fakhouri F, Halimi JM. Etiology and Outcomes of Thrombotic Microangiopathies. Clin J Am Soc Nephrol. 2019 Apr 5;14(4):557-566. doi: 10.2215/CJN.11470918. Epub 2019 Mar 12. PMID 30862697
- [Result] Beczkiewicz ATE, Scharff RL, Kowalcyk BB. Facilitating Evaluation of Hemolytic Uremic Syndrome Long-Term Health Outcomes Through Social Media Support Groups. Front Public Health. 2020 Nov 23;8:544154. doi: 10.3389/fpubh.2020.544154. eCollection 2020. PMID 33330302
- [Result] Alconcher LF, Lucarelli LI, Bronfen S. Long-term kidney outcomes in non-dialyzed children with Shiga-toxin Escherichia coli associated hemolytic uremic syndrome. Pediatr Nephrol. 2023 Jul;38(7):2131-2136. doi: 10.1007/s00467-022-05851-4. Epub 2023 Jan 3. PMID 36595068
- [Result] Ardissino G, Longhi S, Porcaro L, Pintarelli G, Strumbo B, Capone V, Cresseri D, Loffredo G, Tel F, Salardi S, Sgarbanti M, Martelli L, Rodrigues EM, Borsa-Ghiringhelli N, Montini G, Seia M, Cugno M, Carfagna F, Consonni D, Tedeschi S. Risk of Atypical HUS Among Family Members of Patients Carrying Complement Regulatory Gene Abnormality. Kidney Int Rep. 2021 Mar 25;6(6):1614-1621. doi: 10.1016/j.ekir.2021.03.885. eCollection 2021 Jun. PMID 34169201